CLINICAL TRIAL: NCT03558893
Title: Sleep and Circadian Mechanisms Contributing to Nocturnal Non-dipping Blood Pressure
Brief Title: Sleep and Circadian Mechanisms of Non-dipping Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Steven A. Shea, Director, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB 16803
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Hypertension; Cardiovascular Risk Factor
Keywords: circadian rhythm
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Forced Desynchrony (Experimental): All participants will undergo a forced desynchrony protocol.
  Interventions: Behavioral: Forced Desynchrony

INTERVENTIONS:
Behavioral: Forced Desynchrony — All sleep opportunities and other activities will be scheduled by the experimenter so that by the end of the study these activities are spread evenly across all phases of the internal body clock.

SUMMARY:
This study will be the first to distinguish the relative contributions of sleep, circadian and behavioral mechanisms to the non-dipping BP profile in Black adults and will lay the groundwork for optimizing therapies dependent on mechanisms, such as targeting sleep, targeting circadian rhythmicity, or targeting behaviors, and raising the possibility that ideal therapy for hypertension (HTN) may differ by race. This research will ultimately help to improve health and survival in black populations with HTN.

DETAILED DESCRIPTION:
By studying standardized behaviors and regulators of BP during sleep and behavioral stresses across all circadian phases, this protocol will allow us specifically to:

1. To determine if poor sleep, while controlling for circadian phase, contributes to the higher overall BP and reduced nocturnal drop in BP in Blacks compared to Whites.
2. To determine if reduced BP responses to standardized behavioral changes across the day and night contribute to the higher overall BP and reduced nocturnal drop in BP in Blacks compared to Whites.
3. To determine if reduced circadian amplitude of BP contributes to the higher overall BP and reduced nocturnal drop in BP in Blacks compared to Whites.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified Black or White
* 'normotensive' (resting systolic blood pressure (SBP) <140/90 mmHg) or uncomplicated stage 1 'hypertensive' (systolic BP between 140 and 160 mmHg or a diastolic (DBP) between 90 and 100 mmHg).
* free of all prescription and non-prescription drugs (including caffeine, nicotine, alcohol and herbal medications)

Exclusion Criteria:

* Currently treated with pharmacologic agents for hypertension
* Blood pressure >160/100 mmHg
* Smoked within the last year
* Regular night work or rotating shift work for the three months prior to the study
* Travel across more than three time zones during the three months prior to the study.
* Any acute, chronic or debilitating medical conditions, other than mild hypertension (140<SBP<160 or 90<DBP<100 mmHg) and severe renal disease (glomerular filtration rate <30)
* Moderate to severe obstructive sleep apnea (OSA)
* History of severe psychiatric illnesses or psychiatric disorders will be excluded, including alcoholism, drug dependency, major depression, manic depressive illness, schizophrenic disorders, panic disorder, generalized anxiety disorder, post-traumatic stress disorder, agoraphobia, claustrophobia, paranoid personality disorder, schizoid personality disorder, schizotypal personality disorder, borderline personality disorder, and antisocial personality disorder.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 7-day lab stay
  Blood pressure will be measured via automatic and manual-operated sphygmomanometer. Readings will be recorded in units of mmHg.
Heart rate variability | 7-day lab stay
  Two channel ECG will be recorded for heart rate variability analysis.

SECONDARY OUTCOMES:
venous epinephrine | 7-day lab stay
  Venous epinephrine will be measured for adrenal cortex contribution to sympathetic activity.
venous norepinephrine | 7-day lab stay
  venous norepinephrine will be measured for sympathetic nerve activity's contribution to sympathetic activity.
saliva cortisol | 7-day lab stay
  Saliva cortisol will be measured as a sympathetic potentiating hormone.
saliva melatonin | 7-day lab stay
  saliva melatonin will be measured as a sympathetic attenuating hormone.
venous aldosterone | 7-day lab stay
  venous aldosterone will be measured as an end point of renin-angiotensin and sympathetic nerve activation
venous endocannabinoids | 7-day lab stay
  venous endocannabinoids will be measured to estimate stress habituation.
flow mediated dilation | 7-day lab stay
  Flow mediated dilation will be measured as an indication of endothelial function.
beat-by-beat blood pressure | 7-day lab stay
  Beat-by-beat Blood Pressure will be measured in the fingers using a non-invasive blood pressure monitoring device.
24-hr ambulatory blood pressure | 2 day ambulatory period
  Ambulatory blood pressure will be measured with an automatic 24-hr blood pressure monitoring device to estimate of blood pressure dipping status.

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Shea, PhD, Principal Investigator — Ore
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No